CLINICAL TRIAL: NCT01881490
Title: The ImageKids Study: Developing the Pediatric MR Enterography-based Damage Index in Crohn's Disease (pMEDIC) and the Pediatric Inflammatory Crohn's MRE Index (PICMI)
Brief Title: The ImageKids Study: Developing the pMEDIC and the PICMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Collaborators: Children's Hospital of Eastern Ontario (Other); McMaster Children's Hospital (Other); IWK Health Centre (Other); Alberta Children (Unknown); The Hospital for Sick Children (Other); Children's Hospital of Philadelphia (Other); Connecticut Children's Medical Center (Other); Nationwide Children's Hospital (Other); Children's Hospital Medical Center, Cincinnati (Other); Hasbro Children's Hospital (Other); C.S. Mott Children's Hospital (Other); Hospital Sant Joan de Deu (Other); Hospital Materno-Infantil de Málaga (Other); Hôpital Necker-Enfants Malades (Other); Erasmus Medical Center (Other); Leiden University Medical Center (Other); Yorkhill Hospital (Unknown); Dr. von Hauner Children's Hospital (Other); Klinikum Stuttgart (Other); Royal Children's Hospital (Other); Sydney Children's Hospitals Network (Other); Sheba Medical Center (Other Government); Soroka University Medical Center (Other); Rambam Health Care Campus (Other); Schneider Children (Unknown)
Responsible Party: Principal Investigator, Dr Dan Turner, Head of Pediatric Gastroenterology Unit, Shaare Zedek Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ImageKids
Record Dates: First submitted 2013-06-12; First posted 2013-06-19 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; MRE; Pelvic MRI; P-MRI; colonoscopy; gastroscopy
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): 120 Children with Crohn's disease undergoing MRE & colonoscopy will be enrolled and followed for 18 months. MRE exam will be repeated at 18 months.
  Interventions: Device: MRE
- Group 2 (Active Comparator): 120 children with Crohn's disease undergoing colonoscopy will be recruited and will have an MRE/pelvic MRI performed. The two or three contending versions of each index (PICMI and pMEDIC) developed based on Group 1, will be then subjected to head-to-head evaluation of Group 2.
  Interventions: Device: MRE

INTERVENTIONS:
Device: MRE — Developing the Pediatric Crohn's Disease Intestinal Damage Score (pMEDIC score) and the Pediatric MRE-Based Activity Index (PICMI)
  Other Names: MRI; Pelvic MRI

SUMMARY:
The overall objectives of this study are to develop two indices capable of measuring intestinal damage, and, separately, inflammatory disease activity in Pediatric Crohn's disease by means of Magnetic Resonance Imaging with Enterography protocol (MRE) and pelvic MRI.

DETAILED DESCRIPTION:
The PICMI Score and the pMEDIC are aimed to be discriminative (at one point in time), evaluative (measuring damage progression over time) and predictive. The indices will be used as endpoint measures in clinical research and also in clinical practice to identify those who are at risk for rapid disease progression and surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Children (under 18 years of age) with established diagnosis of CD involving any location by the presence of accepted clinical, radiologic, endoscopic and histologic criteria (33, 34).
2. Enrolment at the time of performing ileocolonoscopy and esophageal-gastroduodenoscopy (EGD) as part of clinical care for any reason.
3. Children will be enrolled at any phase of the disease (at diagnosis and thereafter as required clinically). In order to ensure enough subjects with intestinal damage and since damage is progressing over time, enrolment will be stratified based on disease duration. Enrolment for each stratum of disease duration will be closed after reaching the expected sample size.

   * 20% of enrolled children will be within 3 months of diagnosis.
   * 20% of children will be between 3 months and 2 years.
   * 20% will be 2.01 to 3 years
   * 40% will have disease duration over 3-years.
4. Children may be enrolled in any disease activity state (PCDAI 0-100).

Exclusion Criteria:

1. Young children requiring anesthesia for lack of cooperation will be excluded (since the enteric contrast cannot be administered during the 2 hours before anesthesia and it is crucial that the contrast be given just prior the test).
2. For the first 120 children only, subjects not expected to be available for 18 month follow-up, will be excluded (the last 120 subjects may be enrolled as they are not followed longitudinally).

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 240 (Actual)
Dates: Start 2013-01; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Development of MRI-based Index | 3.5 years
  The overall objectives of this study are to develop two indices capable of measuring intestinal damage, and, separately, inflammatory disease activity means of MRE.
  The indices are aimed to be discriminative, evaluative and predictive. they will be used as endpoint measures in clinical research and also in clinical practice to identify those who are at risk for rapid disease progression and surgery. The data collected will be analyzed and scored by both the radiologists and the gastroenterologists. On the basis of these scores, 2 or 3 contending versions of each index will be then subjected to head-to-head evaluation by enrolling another cohort of 120 children undergoing colonoscopy and MRE/pelvic MRI. The best version for each index will be selected according to its performance in the validity, reliability and responsiveness testing. The second group of patients will not be followed longitudinally.

SECONDARY OUTCOMES:
Exploratory | 3.5 years
  To describe the 18-month progression rate of intestinal damage in pediatric Crohn's disease, stratified by the different medications used, and disease duration at enrolment.
Exploratory | 3.5 Years
  To identify biological and clinical markers, predictive of intestinal damage.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Turner, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Derived] Focht G, Cytter-Kuint R, Greer MC, Pratt LT, Castro DA, Church PC, Walters TD, Hyams J, Navon D, Martin de Carpi J, Ruemmele F, Russell RK, Gavish M, Griffiths AM, Turner D. Development, Validation, and Evaluation of the Pediatric Inflammatory Crohn's Magnetic Resonance Enterography Index From the ImageKids Study. Gastroenterology. 2022 Nov;163(5):1306-1320. doi: 10.1053/j.gastro.2022.07.048. Epub 2022 Jul 22. PMID 35872072
- [Derived] Weiss B, Turner D, Griffiths A, Walters T, Herman-Sucharska I, Coppenrath E, Anupindi SA, Towbin AJ, O'Brien K, Silverstein J, Navas V, Koletzko S, Sladek M, Gavish M, Amitai MM; ImageKids study group. NCT01881490. Simple Endoscopic Score of Crohn Disease and Magnetic Resonance Enterography in Children: Report From ImageKids Study. J Pediatr Gastroenterol Nutr. 2019 Oct;69(4):461-465. doi: 10.1097/MPG.0000000000002404. PMID 31136561
- [Derived] Cozijnsen MA, Ben Shoham A, Kang B, Choe BH, Choe YH, Jongsma MME, Russell RK, Ruemmele FM, Escher JC, de Ridder L, Koletzko S, Martin-de-Carpi J, Hyams J, Walters T, Griffiths A, Turner D. Development and Validation of the Mucosal Inflammation Noninvasive Index For Pediatric Crohn's Disease. Clin Gastroenterol Hepatol. 2020 Jan;18(1):133-140.e1. doi: 10.1016/j.cgh.2019.04.012. Epub 2019 Apr 10. PMID 30981008
- [Derived] Weinstein-Nakar I, Focht G, Church P, Walters TD, Abitbol G, Anupindi S, Berteloot L, Hulst JM, Ruemmele F, Lemberg DA, Leach ST, Cytter R, Greer ML, Griffiths AM, Turner D; ImageKids study group. Associations Among Mucosal and Transmural Healing and Fecal Level of Calprotectin in Children With Crohn's Disease. Clin Gastroenterol Hepatol. 2018 Jul;16(7):1089-1097.e4. doi: 10.1016/j.cgh.2018.01.024. Epub 2018 Mar 2. PMID 29501599